CLINICAL TRIAL: NCT05020366
Title: Promoting Health Through Parent Empowerment and the Activation of Routines (Pro-PEAR) Optimization and Feasibility: A Pilot Randomized Controlled Trial (RCT)
Brief Title: Promoting Health Through Parent Empowerment and the Activation of Routines (PrO-PEAR)
Acronym: Pro-PEAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Angela Caldwell, Assistant Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: STUDY21040155; 5K12HD055931-14 (NIH)
Record Dates: First submitted 2021-08-18; First posted 2021-08-25 (Actual); Results first posted 2024-07-15 (Actual); Last update posted 2024-07-15 (Actual); Status verified 2024-06

CONDITIONS: Down Syndrome
Keywords: Early Childhood; Health Promotion; Nutrition; Sleep; Physical Activity
MeSH Terms: conditions — Down Syndrome; Motor Activity

STUDY DESIGN:
Intervention Model Description: Pilot RCT will follow a 2:1 randomization scheme with 2 participant families (parent + child) assigned to intervention (Pro-PEAR) for every 1 assigned to control (enhanced usual care) for a total of 24 participant families.
Who Masked: Outcomes Assessor
Masking Description: Research assistants collecting outcome measures will be blinded to study assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pro-PEAR (Experimental): This group will receive the optimized Pro-PEAR intervention (in addition to usual care).
  Interventions: Behavioral: Promoting Health through Parent Empowerment and the Activation of Routines
- Enhanced Usual Care (Active Comparator): This group will serve as the control group and only receive a report of their child's performance and adherence to World Health Organization recommendations based on baseline data.
  Interventions: Behavioral: Enhanced Usual Care

INTERVENTIONS:
Behavioral: Promoting Health through Parent Empowerment and the Activation of Routines — Parents will receive a report of their child's current performance and adherence to World Health Organization recommendations in each intervention area. Parents will be coached to build consistent family mealtime routines, in which children are involved in meal preparation, food exploration, and play. They will receive education on appropriate serving sizes for young children and basic information nutrition recommendations. Predictable bedtime routines will be designed to incorporate calming sensory input to improve the transition to bed. Parents will be educated on screen time recommendations and help families brainstorm alternatives to screens, including family-based routines of movement and activity. Finally, parents will be coached to incorporate play into all newly adopted routines, as young children learn though play.
  Other Names: Pro-PEAR
  Arms: Pro-PEAR
Behavioral: Enhanced Usual Care — For the control group, usual care will be enhanced by providing parents with a report of their child's performance and adherence to World Health Organization recommendations in the areas of healthy eating, physical activity, sedentary behavior and sleep. This report will consolidate data based on parent report, written logs, and actigraphy at baseline.
  Other Names: EUC
  Arms: Enhanced Usual Care

SUMMARY:
This study will examine the feasibility of the Promoting Health through Parent Empowerment and the Activation of Routines (Pro-PEAR) intervention using a open case-series for intervention optimization followed by a pilot RCT in which participants are randomized to receive Pro-PEAR or enhanced usual care (EUC).

Specific aims include:

1. Optimize the Pro-PEAR intervention manual using an open case series with iterative stakeholder feedback.
2. To determine the feasibility of the Pro-PEAR intervention in terms of recruitment, randomization, retention, adherence, and acceptability.
3. Estimate the effects of the Pro-PEAR intervention on parent reported child health behaviors in each Institute of Medicine obesity prevention area (nutrition, physical activity, sedentary behavior, sleep) over time as compared to a control group.

The following benchmarks will be used to determine feasibility:

Recruitment: >3 parent/child dyads per month Retention: >75% of consented dyads will complete > 8 sessions Adherence: >80% clinician protocol adherence during 100% of sampled sessions Data Collection: >80% planned assessments collected among intervention completers.

Acceptability: >90% of parent intervention completers rate intervention as acceptable.

Additionally, it is predicted that parents will report greater gains in the areas of nutrition, sleep, sedentary behavior and physical activity in the Pro-PEAR group than those in the control group.

DETAILED DESCRIPTION:
Interested participants will contact the research team and screening to determine eligibility may be confirmed in person or over the phone. Interested parent participants will undergo the consent process with a trained research assistant and/or the principal investigator. Families will be sent the informed consent documents prior to informed consent process. Prior to data collection, a member of the research team will use a script to discuss the risks and activities involved in study participation and answer any questions the participant has about the study. Following signed informed consent, an appointment will be scheduled for baseline assessments.

Child participants will be provided with the wrist-worn actigraphy device and thigh-worn Physical Activities Logging (activPAL) device, and parents/caregivers educated on the wear schedule and periodic skin checks to ensure skin integrity. Parents will be instructed to complete skin checks daily to minimize risk of abrasions and to contact the study team immediately if any issues occur. The child will wear these devices to collect data on activity, sedentary behavior, and sleep for 7 full days. It is anticipated that each assessment appointment will last approximately 2 hours. If conducted remotely, devices and other materials will be mailed to the participant and completed with a member of the research team on the phone or video conference to answer any question. Equipment will be collected at the time of the first in- person intervention session or by placing in a pre-paid postage box (provided by research team) and placing in the mail.

After assessments, the first approximately ten families will receive the Pro-PEAR intervention from Caldwell (PI) over 12 sessions in their home. Every other week (weeks: 1, 3, 5, 7, 9, 11) parents will be coached on a new health promoting topic: family meals, healthy portions, bedtime routines, strategies for screens, moving and grooving, and health promoting play. Each of these sessions will last approximately 30 minutes and may be delivered in person or remotely (using Zoom). During the alternate weeks (2, 4, 6, 8, 10, 12) therapists will check in with families and address any issues or barriers (such as child behavior) that has impacted progress toward building healthy habits. Each of these sessions will last approximately 30 minutes and be delivered remotely via Zoom.

Data collected from these first ~10 families will inform intervention optimization and finalization of the manual of procedures for the pilot RCT. Once the manual is finalized, 24 additional families will be recruited and randomized (2:1) to receive either Pro-PEAR or a control (enhanced usual care). Families assigned to Pro-PEAR will receive intervention as described above with minor modification as informed by the first 10 participants. Pro-PEAR will be delivered by trained occupational therapy clinicians. Families assigned to control will receive enhanced usual care. Enhanced usual care will include information about child habits in the areas of healthy eating, physical activity, sedentary behavior and sleep based on parent questionnaires and actigraphy. For both the Pro-PEAR and the control group, usual care will be documented through questions about receipt of services and semi-structured interviews with parents.

Parent Experience:

All research activities will take place in the participants' homes. Parents will be expected to complete assessment and intervention activities in the comfort of their home with the research team joining in-person or virtually as needed/preferred. They may refuse to participate in any portion of the research study at any time and will be encouraged to be an active collaborator throughout all actives.

Child Experience:

Children will be expected to wear the Phillips Actiwatch on their wrist and the activPAL on their thigh for 1 week at each assessment timepoint. Children will be expected to participate in activities initiated by their parents and clinicians as appropriate throughout all phases of research.

Based on prior studies within the lab, it is anticipated that >75% of participants will complete the 3-month program and 6 month follow-up (>18/24). A sample size of 24 in the pilot RCT will provide us with the >12 PrO-PEAR intervention completers needed to estimate average outcome values and variability to plan larger subsequent trials.

Descriptive statistics will be used to determine whether feasibility benchmarks have been met for each group. Between group differences and differences in primary outcomes over time will be analyzed using linear mixed models with fixed and random effects.

ELIGIBILITY:
Child Inclusion Criteria:

1. between the ages of 12 and 36 months
2. diagnosis of Down syndrome
3. demonstrate independent mobility (e.g., walking, crawling)

Child Exclusion Criteria:

1. mobility is significantly restricted because of a medical condition, or
2. nutrition is received primarily by feeding tube.

Parent Inclusion Criteria

1) aged > 18 years

Parent Exclusion Criteria

* N/A

Min Age: 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-10-04 (Actual); Primary Completion 2023-05-23 (Actual); Study Completion 2023-05-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Angela Caldwell, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- Down Syndrome Center of Western Pennsylvania, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
There are currently no plans to share individual participant data. Individual participant data will be shared with other researchers upon reasonable request and with approved data use agreement in place.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Protocol Enrollment reflects the number of individual children and parents enrolled [40], but data are reported in the Results Section per family unit [20], except where otherwise noted [Adverse Events].
Period: Overall Study
Arm/Group | Pro-PEAR | Enhanced Usual Care
Started | 15 | 5
Completed | 11 | 5
Not Completed | 4 | 0
Not completed — Lost to Follow-up | 2 | 0
Not completed — Withdrawal by Subject | 2 | 0

BASELINE CHARACTERISTICS:
Population: We collected baseline measures on 20 child participants that are included in the baseline analysis.
Groups:
- Pro-PEAR: This group will receive the optimized Pro-PEAR intervention (in addition to usual care).
  Parents will receive a report of their child's current performance and adherence to World Health Organization recommendations in each intervention area. Parents will be coached to build consistent family mealtime routines, in which children are involved in meal preparation, food exploration, and play. They will receive education on appropriate serving sizes for young children and basic information nutrition recommendations. Predictable bedtime routines will be designed to incorporate calming sensory input to improve the transition to bed. Parents will be educated on screen time recommendations and help families brainstorm alternatives to screens, including family-based routines of movement and activity. Finally, parents will be coached to incorporate play into all newly adopted routines, as young children learn though play.
- Total: Total of all reporting groups
Arm/Group | Pro-PEAR | Enhanced Usual Care | Total
Number analyzed (Participants) | 15 | 5 | 20
Age, Continuous [Mean (Standard Deviation); unit: months] — Children
  months | 26.1 (7.4) | 30.2 (6.0) | 27.2 (7.2)
Age, Continuous [Mean (Standard Deviation); unit: years] — Parents Population: Two parents did not provide age data. Only those with age data were included in this report.
  years
    number analyzed (Participants) | 13 | 5 | 18
    (all) | 35.6 (3.7) | 34.4 (6.0) | 35.2 (4.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Child Participants: Female | 6 | 2 | 8
  Child Participants: Male | 9 | 3 | 12
  Parent Participants: Female | 14 | 5 | 19
  Parent Participants: Male | 1 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Child Participants: Hispanic or Latino | 2 | 1 | 3
  Child Participants: Not Hispanic or Latino | 13 | 4 | 17
  Child Participants: Unknown or Not Reported | 0 | 0 | 0
  Parent Participants: Hispanic or Latino | 1 | 1 | 2
  Parent Participants: Not Hispanic or Latino | 14 | 4 | 18
  Parent Participants: Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  Child Participants: American Indian or Alaska Native | 0 | 0 | 0
  Child Participants: Asian | 0 | 0 | 0
  Child Participants: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Child Participants: Black or African American | 2 | 0 | 2
  Child Participants: White | 9 | 5 | 14
  Child Participants: More than one race | 3 | 0 | 3
  Child Participants: Unknown or Not Reported | 1 | 0 | 1
  Parent Participants: American Indian or Alaska Native | 0 | 0 | 0
  Parent Participants: Asian | 0 | 0 | 0
  Parent Participants: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Parent Participants: Black or African American | 1 | 0 | 1
  Parent Participants: White | 12 | 5 | 17
  Parent Participants: More than one race | 0 | 0 | 0
  Parent Participants: Unknown or Not Reported | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Pro-PEAR Intervention Sessions Completed
Description: As measured using interventionist documentation
Time Frame: 3 months
Population: In this analysis, we only included participants (both children and parents) who attended at least 1 intervention session (e.g., not those lost to follow-up prior to intervention and not those in the control group.
Measure: Mean (Standard Deviation); unit: # of sessions completed
Arm/Group | Pro-PEAR | Enhanced Usual Care
Number analyzed (Participants) | 14 | 0
# of sessions completed | 9.1 (2.3) |

2. Primary Outcome: Parent-reported Intervention Acceptability as Rated on a Likert Scale.
Description: Participant acceptability ratings of the PrO-PEAR intervention using the Treatment Acceptability Questionnaire. Scores range from 8 to 48 with higher scores indicating higher acceptability.
Time Frame: 3 months
Population: The TAQ was sent separately only to parent participants who received the intervention. Not all parent participants who received this web-based survey completed it.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Pro-PEAR | Enhanced Usual Care
Number analyzed (Participants) | 8 | 0
score on a scale | 38.8 (6.8) |

3. Primary Outcome: Percentage of Planned Data Collection Efforts Completed Successfully
Description: Measured by the number of outcomes collected divided by the number of planned outcomes
Time Frame: 6 months
Population: We calculated the number of outcomes collected across participants in the intervention and control groups and calculated percentage of assessments collected.
Measure: Number; unit: percentage of assessments collected
Units Other Than Participants: Planned Assessments
Arm/Group | Pro-PEAR | Enhanced Usual Care
Number analyzed (Participants) | 15 | 5
Number analyzed (Planned Assessments) | 450 | 150
percentage of assessments collected | 80 | 94

4. Primary Outcome: Number of Participant Families Recruited Per Month
Description: Quantified for each month of active recruitment and averaged
Time Frame: up to 1 year
Population: Participant families were randomized to groups after recruitment - we report this data based on family units.
Measure: Number; unit: participant families per month
Groups:
- Trial Recruitment: Participants were recruited prior to randomization into groups
Arm/Group | Trial Recruitment
Number analyzed (Participants) | 20
participant families per month | 5.25

5. Secondary Outcome: Change in Healthy Eating From Baseline to 3 Months
Description: change in # of fruits & vegetables children consumed, on average, each day as measured by parent report and the EAT FFQ (Eating Assessment in Toddlers Food Frequency Questionnaire).
  Average number of portions of fruits and vegetables were reported on two questions of a Food Frequency Questionnaire with options ranging from 0-4 servings of fruits and 0-4 servings of vegetables. These scores were added together at each time point with greater scores indicating greater consumption of fruits and vegetables.
Time Frame: baseline to 3 months
Population: We only used outcomes on child participants with complete data at baseline and 3 months.
Measure: Mean (Standard Deviation); unit: change score on a scale
Arm/Group | Pro-PEAR | Enhanced Usual Care
Number analyzed (Participants) | 12 | 5
change score on a scale | 0.33 (1.03) | 0.2 (1.17)

6. Secondary Outcome: Change in Healthy Eating From Baseline to 6 Months
Description: as for outcome 5
Time Frame: baseline to 6 months
Population: We only analyzed child participants with complete data at baseline and 6 months on this measure.
Measure: Mean (Standard Deviation); unit: change score on a scale
Arm/Group | Pro-PEAR | Enhanced Usual Care
Number analyzed (Participants) | 9 | 5
change score on a scale | 0.11 (1.52) | -0.2 (1.17)

7. Secondary Outcome: Change in Physical Activity From Baseline to 3 Months
Description: change in # of hours of light, moderate, or vigorous child physical activity, on average, each day as measured by activPAL
Time Frame: baseline to 3 months
Population: We only analyzed data on child participants with data on physical activity at baseline and 3 months.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Pro-PEAR | Enhanced Usual Care
Number analyzed (Participants) | 9 | 3
hours | 0.45 (1.97) | 0.01 (0.78)

8. Secondary Outcome: Change in Physical Activity From Baseline to 6 Months
Description: as for outcome 7
Time Frame: baseline to 6 months
Population: We only analyzed data on child participants with complete physical activity data at baseline and 6 months.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Pro-PEAR | Enhanced Usual Care
Number analyzed (Participants) | 8 | 4
hours | 0.32 (1.35) | 1.33 (0.89)

9. Secondary Outcome: Change in Sedentary Behavior From Baseline to 3 Months
Description: change in # of minutes spent in bouts of sedentary behavior >60 minutes, on average, each day as measured by activPAL (Physical Activities Logging)
Time Frame: baseline to 3 months
Population: Only child participants with complete data for sedentary behavior (activPAL) at baseline and 3 months were included.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Pro-PEAR | Enhanced Usual Care
Number analyzed (Participants) | 8 | 3
minutes | 21.01 (73.35) | 11.66 (31.93)

10. Secondary Outcome: Change in Sedentary Behavior From Baseline to 6 Months
Description: change in # minutes of bouts of sedentary behavior >60 minutes, on average, each day as measured by activPAL
Time Frame: baseline to 6 months
Population: Only child participants with complete data for sedentary behavior (activPAL) at baseline and 6 months were included.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Pro-PEAR | Enhanced Usual Care
Number analyzed (Participants) | 7 | 3
minutes | -32.54 (70.52) | -54.45 (38.16)

11. Secondary Outcome: Change in Sleep Duration From Baseline to 3 Months
Description: change in # minutes of child sleep, on average, each night as measured by the Phillips Actiwatch
Time Frame: baseline to 3 months
Population: We only included child participants with data for sleep (Actiwatch) at baseline and 3 months.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Pro-PEAR | Enhanced Usual Care
Number analyzed (Participants) | 11 | 5
minutes | 13.50 (50.03) | 9.68 (34.00)

12. Secondary Outcome: Change in Sleep Duration From Baseline to 6 Months
Description: change in # minutes of child sleep, on average, each night as measured by the Phillips Actiwatch
Time Frame: baseline to 6 months
Population: Only child participants who had sleep (Actiwatch) data at baseline and 6 months were included.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Pro-PEAR | Enhanced Usual Care
Number analyzed (Participants) | 8 | 5
minutes | 19.26 (52.02) | 21.12 (18.11)

13. Secondary Outcome: Change in Child Weight From Baseline to 6 Months
Description: Child weight will be assessed using chart review and scale
Time Frame: baseline to 6 months
Population: We only analyzed child participants with complete data on weight at baseline and 6 months.
Measure: Mean (Standard Deviation); unit: pounds
Arm/Group | Pro-PEAR | Enhanced Usual Care
Number analyzed (Participants) | 9 | 5
pounds | 4.40 (0.74) | 3.38 (0.99)

14. Secondary Outcome: Change in Child Height From Baseline to 6 Months
Description: Child weight will be assessed using chart review and scale
Time Frame: baseline to 6 months
Population: We only analyzed child participants with complete height data at baseline and 6 months.
Measure: Mean (Standard Deviation); unit: inches
Arm/Group | Pro-PEAR | Enhanced Usual Care
Number analyzed (Participants) | 9 | 3
inches | 3.78 (4.13) | 4.84 (2.64)

15. Secondary Outcome: Change in Child Weight From Baseline to 1 Year
Description: Child weight will be assessed using chart review.
Time Frame: 1 year
Population: We were unable to collect this data because we could not gain access to participant's charts throughout the conduct of this study.
Arm/Group | Pro-PEAR | Enhanced Usual Care
Number analyzed (Participants) | 0 | 0

16. Secondary Outcome: Change in Child Height From Baseline to 1 Year
Description: Child height will be assessed using chart review.
Time Frame: one year
Population: We were unable to collect height at one year because we were not able to gain access to participant's medical chart throughout the conduct of this study.
Arm/Group | Pro-PEAR | Enhanced Usual Care
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 6 months
Description: Participants were encouraged to report adverse events experienced as part of data collection. We are reporting on adverse events reported for child and parent participants.
Groups:
- PrO-PEAR: This group will receive the optimized PrO-PEAR intervention (in addition to usual care).
  Preventing Obesity through Parent Empowerment and the Activation of Routines: Parents will receive a report of their child's current performance and adherence to World Health Organization recommendations in each intervention area. Parents will be coached to build consistent family mealtime routines, in which children are involved in meal preparation, food exploration, and play. They will receive education on appropriate serving sizes for young children and basic information nutrition recommendations. Predictable bedtime routines will be designed to incorporate calming sensory input to improve the transition to bed. Parents will be educated on screen time recommendations and help families brainstorm alternatives to screens, including family-based routines of movement and activity. Finally, parents will be coached to incorporate play into all newly adopted routines, as young children learn though play.
Arm/Group | PrO-PEAR | Enhanced Usual Care
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/10
Other Adverse Events (participants affected / at risk) | 1/30 | 0/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PrO-PEAR (N=30) | Enhanced Usual Care (N=10)
skin irritation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Skin irritation (redness) is caused by the application of an activPAL device to the thigh with medical tape.

LIMITATIONS AND CAVEATS:
This trial's limitations include a small sample size and a 2:1 randomization scheme, which gives preference to the intervention group due to this being a feasibility study. Therefore, group comparisons would not be meaningful.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-12-12): https://cdn.clinicaltrials.gov/large-docs/66/NCT05020366/Prot_SAP_001.pdf
  • Informed Consent Form (2022-12-12): https://cdn.clinicaltrials.gov/large-docs/66/NCT05020366/ICF_000.pdf